CLINICAL TRIAL: NCT06790095
Title: Transforming Research and Clinical Knowledge in Traumatic Brain Injury (TRACK-TBI) Precision Medicine Part 3 - Option II
Brief Title: TRACK-TBI Precision Medicine Part 3 - Option II
Acronym: PM-003
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PM-003
Record Dates: First submitted 2025-01-17; First posted 2025-01-23 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Cyclosporine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cyclosporine (CsA) (Active Comparator): Intravenous (IV) injection, 2.5 mg/kg loading dose given over 2 hours, followed by a 3-day (72-hour) constant IV infusion of 5 mg/kg/day.
  Interventions: Drug: Cyclosporine (CsA)
- Matching Placebo (Placebo Comparator): Intravenous (IV) injection of 0.9% NaCl over 74 hours.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cyclosporine (CsA) — Intravenous (IV) injection, loading dose of 2.5 mg/kg (diluted in 0.9% NaCl to a final volume of 50 ml) given over 2 hours, immediately followed by a continuous IV infusion of of 5 mg/kg/day (diluted in 0.9% NaCl to a final volume of 250 ml) for 3 days (72-hour).
  Other Names: Sandimmune®
  Arms: Cyclosporine (CsA)
Drug: Placebo — Intravenous (IV) injection of 0.9% NaCl with the same dosing strategy as CsA: "loading dose" given over 2 hours, immediately followed by a continuous IV infusion for 3 days (72-hour).
  Arms: Matching Placebo

SUMMARY:
The purpose of this study is to determine if experimental drug treatment improves recovery after TBI as compared to a control (placebo) group. Changes in recovery will be measured throughout the study. The study drug listed below is approved by the U.S. Food and Drug Administration (FDA) but is being used "off-label" in this study. This means that the drug is not currently approved to treat TBI.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (18-65 years of age, inclusive)
2. Presents to a participating enrollment site and is able to receive treatment within 24 hours of head injury warranting clinical evaluation with a non- contrast cranial CT based on American College of Emergency Physicians (ACEP) Centers for Disease Control and Prevention (CDC) clinical policy for TBI imaging.
3. Closest, prior to randomization GCS score of 3 to 8
4. Evidence of TBI on cranial CT, confirmed by:

   * Evidence of contusion and/or
   * Evidence of traumatic axonal microvascular injury (TAMVI)
5. Initial GFAP blood level >1000 pg/mL ≤ 15000 pg/mL determined using a for Research Use Only (RUO) assay(s) or an Investigation Use Only (IUO) assay(s)
6. Participants able to undergo Magnetic Resonance Imaging (MRI) scans, no contraindications
7. Legally Authorized Representative (LAR) willing and able to provide informed consent
8. Participant/LAR able to read, speak, and understand English or Spanish (participating site dependent, where available), including the Informed Consent Form (ICF)

Exclusion Criteria:

1. Isolated epidural hematoma
2. Bilaterally fixed dilated pupils in the absence of paralytic medications, or evidence of herniation on cranial CT
3. Pre-existing conditions including disabling developmental, neurologic, psychiatric, medical disorder that continues to produce functional disability up to the time of injury; or imminent death based on clinical judgement
4. Order for comfort care placed prior to enrollment
5. Current enrollment in another interventional study
6. Currently pregnant or currently breastfeeding or planning on becoming pregnant in the next 6M
7. Current incarceration or in custody
8. On psychiatric hold (e.g. Codes 5150, 5250)
9. Ongoing pre-injury therapy with the Investigational Product (IP), currently receiving immunosuppressive therapy or any contraindicated medications (see CsA Drug contraindications/caution table in Manual of Procedures)
10. Current or medical history of any allergic reactions and/or anaphylactic reactions towards CsA and cremophor (also known as kolliphor®)
11. Severe polytrauma or previous conditions that would preclude conducting any study activities
12. Any spinal cord injury of grade A to D on the American Spinal Injury Association (ASIA) Impairment Scale
13. Primary diagnosis at the enrolling facility of ischemic or hemorrhagic stroke
14. Body Mass Index (BMI) >35
15. Hemodynamic instability, per participating site physician investigator clinical judgement
16. Current or medical history of renal dysfunction, significant renal failure, or high-risk for renal failure, defined as:

    * Creatinine Clearance (CrCl) or estimated Glomerular Filtration Rate (eGFR) (<60 mL/minute/1.73 m2)
    * Major rhabdomyolysis with creatine kinase > 5,000 IU/L
17. Current or medical history of hepatic disease or serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) value >3 times the upper limit of normal lab value at the screening/baseline visit
18. Current or medical history of serious chronic viral or fungal infection
19. Current or medical history of active mycobacterial infection or anti- tuberculous treatment
20. Medical history of human immunodeficiency virus, hepatitis B surface antigen, or hepatitis C virus antibody
21. Any significant disease or disorder (including abnormal laboratory tests) which, in the opinion of the participating site investigator, may either put the patient at risk because of participation in the study, or may influence the results of the study
22. Low likelihood of follow up or study compliance, or any other reason, in the opinion of the participating site investigator, the participants should not participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Change in Disability Rating Score (DRS) | Baseline to Week 4 post-injury
  The primary outcome measure is to determine whether the intervention safely improves functional outcome in participants with TBI as compared to placebo, as measured by the change in the Disability Rating Score (DRS) score from Baseline to Week 4 post-injury.

SECONDARY OUTCOMES:
Change in Blood-based biomarker (Neurofilament light chain) | Baseline to Week 2 post-injury
  To determine whether the intervention lowers the rising plasma Neurofilament light chain (NfL) levels up to W2 post-injury in participants with TBI as compared to placebo.
Change in Blood-based biomarker (GFAP) | Baseline to Week 2 post-injury
  To determine whether the intervention lowers the plasma GFAP levels up to W2 post-injury as compared to placebo.
Change in Blood-based biomarker (UCH-L1) | Baseline to Week 2 post-injury
  To determine whether the intervention lowers the plasma UCH-L1 levels up to Week 2 post-injury in participants with TBI as completed to placebo.
Post-TBI symptom outcome (CRSR-FAST) | Baseline to Week 4 post-injury
  To determine the effect of intervention on the change in the number of behavioral signs of consciousness present on the Coma Recovery Scale- Revised For Accelerated Standardized Testing (CRSR-FAST) from Baseline to W4 post-injury as compared to placebo.
Imaging biomarkers | Week 2 to Month 6
  To determine whether the intervention results in improved imaging biomarkers compared to placebo measured by: 1) the change in white matter tract using MRI diffusion tensor imaging (DTI), and 2) change in total brain volumetrics using MRI T1 MPRAGE, from Week 2 to Month 6.
Post-TBI functional outcomes (DRS) | Baseline to Month 3 and Baseline to Month 6
  To determine the effect of intervention on functional outcomes, as measured by:
  I. Change in the Disability Rating Scale (DRS) from Baseline to Month 3 and Baseline to Month 6
Post-TBI functional outcomes (FSE) | Week 2, Week 4, Month 3 and Month 6
  To determine the effect of intervention on functional outcomes, as measured by:
  II. Functional Status Examination (FSE) score at Week 2, Week 4, Month 3 and Month 6
Post-TBI functional outcomes (GOSE-TBI) | Week 2, Week 4, Month 3 and Month 6
  To determine the effect of intervention on functional outcomes, as measured by:
  III. Glasgow Outcome Scale Extended (TBI Version) (GOSE-TBI) score at Week 2, Week 4, Month 3 and Month 6.
Post-TBI cognitive outcome (BTACT) | Week 4, Month 3, and Month 6
  To determine the effect of the intervention on cognitive outcome, as measured by the Brief Test of Adult Cognition by Telephone (BTACT) Composite z-score at Week 4, Month 3 and Month 6.
Post-TBI quality of life and patient-reported outcomes (QOLIBRI) | Month 3 and Month 6
  To determine the effect of intervention on quality of life and other patient-reported outcomes (PRO), as measured by the Quality of Life Brain Injury (QOLIBRI) at Month 3 and Month 6.
Post-TBI quality of life and patient-reported outcomes (RPQ) | Month 3 and Month 6
  To determine the effect of intervention on quality of life and other patient-reported outcomes (PRO), as measured by the Rivermead Post Concussion Symptoms Questionnaire (RPQ) at Month 3 and Month 6.
Post-TBI quality of life and patient-reported outcomes (Caregiver Burden) | Month 3 and Month 6
  To determine the effect of intervention on quality of life and other patient-reported outcomes (PRO), as measured by the Caregiver Burden at Month 3 and Month 6.

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Manley, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available through the Federal Interagency TBI Research (FITBIR) Database.
Time Frame: Shared scientific data will be made accessible as soon as possible, and no later than the time of an associated publication, or the end of performance period, whichever comes first.
Access Criteria: FITBIR qualified investigators will be provided access
URL: https://fitbir.nih.gov/

REFERENCES:
- See also: Related Info — https://tracktbi.ucsf.edu/
- See also: Related Info — https://tracktbi.ucsf.edu/publications
- See also: Related Info — https://tracktbinet.ucsf.edu/